CLINICAL TRIAL: NCT04881513
Title: The Structure and the Function of the Taste Buds After the Stapes Surgery and the Patients Quality of Life and it's Correlation to the Change of the Threshold of the Chorda Tympani Electrical Stimulation
Brief Title: The Change of the Structure and Function of Taste Buds After the Otosclerosis Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Nina Bozanic Urbancic, MD, ENT specialist, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHORDA_TASTE_OTOSCLEROSIS
Record Dates: First submitted 2021-01-07; First posted 2021-05-11 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Chorda Tympani Disorder; Taste Disorders; Stapes Fixation
Keywords: stapedectomy; taste; taste buds; chorda tympani; narrow band imaging; electrical stimulation; taste strips; two point discrimination; quality of life
MeSH Terms: conditions — Taste Disorders | interventions — Narrow Band Imaging; Taste

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Structure /function of the taste buds and QoL (Other): The structure of the taste buds is measured by Narrow Band Imaging (NBI) technique prior to the operation, one month and six months after the surgery.
  The tongue sensation is measured by two point discrimination before the operation, one month and six months after the operation.
  The taste is tested by the taste strips prior to, on month and six month after the surgery.
  The quality of life is measured by the SF36 questionnaire. The threshold change is measured by the stimulating electrode at the beginning and at the end of the surgery.
  Interventions: Diagnostic Test: Narrow Band Imaging; Diagnostic Test: Tongue sensitivity testing; Other: Qualitiy of life; Diagnostic Test: Threshold change; Diagnostic Test: Taste

INTERVENTIONS:
Diagnostic Test: Narrow Band Imaging — Testing the taste buds structure (blood vessels morphology- classified to 5 types) and the number of taste buds per 20mm2, by Narrow Band Imaging technique before and after the operation (one and six months)
  Other Names: NBI
Diagnostic Test: Tongue sensitivity testing — testing the tongue sensitivity change prior to surgery and after (1 and 6 months) the surgery with two point discrimination test in mm.
  Other Names: Two point discriminator
Other: Qualitiy of life — Testing the patients quality of life before and after (one and six months) the stapes surgery by SF 36 questionnaire
  Other Names: SF36
Diagnostic Test: Threshold change — Measuring the intraoperative chorda tympani stimulation threshold change at the beginning and at the end of the procedure- surgery
Diagnostic Test: Taste — Taste is measured by applying taste strips (sweet, sour, salty, bitter) in 4 concentrations prior to, 1 and 6 months after surgery.

SUMMARY:
Patients admitted for the otosclerosis operation are included in the study. The Narrow Band Imaging (NBI) of their taste buds is performed before the operation. The sensory function of the anterior 2/3 of the tongue is tested with the two point discrimination discs, the taste is tested with taste strips and the SF-36 questionnaire is applied. During the operation in local anesthesia the threshold for the tongue sensation (by the stimulation of the chorda tympani nerve) of the first 2/3 of the tongue at the beginning of the operation (when we first encounter the chorda tympani nerve) and at the end of the operation is measured.One month and six months after the operation the tests are being repeated (NBI, two-point discrimination and SF-36 questionnaire).

The study has the National Ethical Committee approval.

DETAILED DESCRIPTION:
Patients admitted for otosclerosis operation 18 to 65 years old, not taking medications that could influence the taste and not having the problems with the smell are being recruited for the study.

The informed consent is signed by the patient. The Narrow Band Imaging (NBI) of their taste buds is performed before the operation. The number of taste buds in the 20mm2 size area and the blood vessel morphology is being recorded. For the blood vessel morphology the five point scoring system is used. Both sides of the tongue are tested separately.

The sensory function of the anterior 2/3 of the tongue is tested with the two point discrimination discs. Both sides of the tongue are tested separately.

The taste strips are used with 4 different concentrations of sweet, sour, salty and bitter applied to each side of the tongue separately.

SF-36 questionnaire adapted to Slovenian language is applied. During the operation in local anesthesia the threshold for the tongue sensation at the beginning of the operation (when the investigators first encounter the chorda tympani nerve) and at the end of the operation is measured. The investigators use the facial nerve monitoring system for the measurements and stimulate directly the chorda tympani with electrical current. After each operation the surgeon determines the grade of the intraoperative manipulation of the chorda tympani nerve.

One month and six months after the operation the tests are being repeated (NBI, two-point discrimination, taste testing with taste strips and SF-36 questionnaire).

The study has the National Ethical Committee approval.

ELIGIBILITY:
Inclusion Criteria: otosclerosis surgery -

Exclusion Criteria: smell disturbance, taking drugs that could have the influence on taste, diseases and injuries of the tongue

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The change of the count of the taste buds after stapes surgery mesured by NBI | 2 years
  The evaluation of the influence of the manipulation of the chorda tympani nerve on the structure of the taste buds measured by Narrow Band Imaging technique prior to surgery and 1 month and 6 months after surgery. The number of the taste buds will be counted on the surface of 20 mm2 .
The change of the structure -blood vessel morphology of the taste buds after stapes surgery mesured by NBI | 2 years
  The evaluation of the influence of the manipulation of the chorda tympani nerve on the structure of the taste buds measured by Narrow Band Imaging technique prior to surgery and 1 month and 6 months after surgery. The blood vessel morphology will be assessed by the 5-point scoring system.
The change of the function of the taste buds mesured by the test strips | 2 years
  The evaluation of the influence of the chorda tympani intraoperative manipulation to the change of the chorda tympani function measured by the taste strips test.
The influence of the chorda tympani intraoperative manipulation on the patients quality of life | 2 years
  The patients quality of life is measured by the SF 36 questionnaire
The change of the function of the chorda tympani nerve measured by the change of tongue sensitivity measured by two point discrimination test | 2 years
  The evaluation of the influence of the chorda tympani intraoperative manipulation to the change of the chorda tympani function measured by the two pint dicrimination test ( in mm)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Božanić Urbančič, MD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No